CLINICAL TRIAL: NCT00514982
Title: An Observational Study of the Immunopathogenesis of and Response to Step-Up Inflammatory Bowel Disease Therapy for Hermansky-Pudlak Syndrome-Associated Colitis
Brief Title: Medical Treatment of Colitis in Patients With Hermansky-Pudlak Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Michael D. Yao, M.D./National Institute of Allergy and Infectious Diseases, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070205; 07-I-0205
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-03-08

CONDITIONS: Hermanski-Pudlak Syndrome; Colitis; Cytokines; Lymphocytes; Drug Evaluation
Keywords: Hermansky-Pudlak Syndrome; Colitis; Medical Therapy; Immunopathogenesis; Cytokine; Hermansky-Pudlak Syndrome Associated Colitis; HPS
MeSH Terms: conditions — Hermanski-Pudlak Syndrome; Colitis | interventions — Mesalamine; Infliximab; Adrenal Cortex Hormones; Mercaptopurine; Tacrolimus; Adalimumab

ARMS (6):
- 1/Drug #1 (Other): Oral mesalamine will be used as initial therapy in patients who are not taking any medication or have not received any prior treatment for their IBD. Dosing will begin at 2.4 g PO QD and will be increased to 4.8 g QD within 2 weeks. Topical mesalamine (enema 4 g PR HS/BID or suppository 1 g PR HS/BID) may be added for patients with inflammation that is limited to the rectum (proctitis) or who have prominent complaints of urgency, incomplete evacuation or rectal bleeding.
  Interventions: Drug: Mesalamine
- 1/Drug#2 (Other): Add oral corticosteroids (prednisone) to mesalamine. The standard induction dose will be 40 mg/day. After 1 week of therapy, if the total SCCAI score has decreased by greater than or equal to 2 points the patient will continue on another week of therapy. If the SCCAI has not decreased by greater than or equal to 2 points (indicative of a reduction in symptoms) at one week, then the dose will be increased to 60 mg/day. Patients on either dosage will have another SCCAI assessment done a week later (2 weeks after beginning corticosteroids), and if they are found to be in remission (SCCAI less than or equal to 2), a steroid-tapering schedule will be initiated.
  Interventions: Drug: Corticosteroids
- 1/Drug#3 (Other): Infliximab and 6-MP will be added to patients with a SCCAI greater than 2 at week 8. The first infusion of infliximab (5 mg/kg) will be given during that week. In addition, 6-MP will be initiated at doses of 1.0-1.5 mg/kg PO QD to reduce the incidence of infliximab antibody formation and facilitate steroid tapering (the target dose of 6-MP will be decreased accordingly if patients are found to have low TMPT levels/activity by genotypic or phenotypic testing). Also, steroids will also be rapidly tapered off at this time.
  Interventions: Drug: 6-Mercaptopurine
- 1/Drug#4 (Other): Infliximab and 6-MP will be added to patients with a SCCAI greater than 2 at week 8. The first infusion of infliximab (5 mg/kg) will be given during that week. In addition, 6-MP will be initiated at doses of 1.0-1.5 mg/kg PO QD to reduce the incidence of infliximab antibody formation and facilitate steroid tapering (the target dose of 6-MP will be decreased accordingly if patients are found to have low TMPT levels/activity by genotypic or phenotypic testing). Also, steroids will also be rapidly tapered off at this time.
  Interventions: Drug: Infliximab
- 1/Drug#5 (Other): Subjects with a SCCAI greater than 2 after 3 doses of infliximab will continue 6-MP, discontinue infliximab infusions and start adalimumab injections approximately 2 weeks after the 3rd dose of infliximab. Induction dosing will consist of a 160 Micro/g subcutaneous injection, followed by 80 Micro/g 2 weeks after.
  Interventions: Drug: Adalimumab
- 1/Drug#6 (Other): Patients who have a SCCAI greater than 2 after 2 doses of adalimumab will continue 6-MP, discontinue adalimumab, and start therapy with tacrolimus 0.01 mg/kg PO BID approximately 2 weeks after the second dose of adalimumab.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Mesalamine — 5-Aminosalicylic Acid Derivative used to treat mild to moderate Ulcerative Colitis
  Arms: 1/Drug #1
Drug: Infliximab — Antirheumatic, Disease Modifying Gastrointestinal Agent, Miscellaneous, Monoclonal Antibody, Tumor Necrosis Factor (TNF) Blocking Agent used to treat gastrointestinal disorders.
  Arms: 1/Drug#4
Drug: Corticosteroids — Systemic Corticosteroid used to treat inflammatory conditions.
  Arms: 1/Drug#2
Drug: 6-Mercaptopurine — Antineoplastic Agent, Antimetabolite, Immunosuppressant Agent used traditionally to treat Acute lymphoblastic leukemia. Unlabeled use as steroid-sparing agent for corticosteroid-dependent Crohn's disease (CD) and ulcerative colitis (UC); maintenance of remission in CD; fistulizing Crohn's disease.
  Arms: 1/Drug#3
Drug: Tacrolimus — Immunosuppressant Agent used to treat Liver, Heart, Kidney transplant, prevent host vs graft disease, severe atopic dermatitis.
  Arms: 1/Drug#6
Drug: Adalimumab — Antirheumatic, Monoclonal Antibody, Tumor Necrosis Factor (TNF) Blocking Agent used to treat Rheumatoid arthritis and Crohn's disease.
  Arms: 1/Drug#5

SUMMARY:
This study will determine if medical treatment of colitis (inflammation of the colon resulting in loose bowel movements, rectal bleeding, and belly pain) that is used for other colitis conditions, such as Crohn's disease and ulcerative colitis, is safe and effective for treating colitis in patients with Hermansky-Pudlak syndrome (HPS). HPS is a hereditary disorder that causes albinism, visual impairment, and abnormal bleeding. Some patients also develop colitis, pulmonary fibrosis, and kidney disease.

Patients with HPS and colitis who are 18 years of age or older may be eligible for this study. Participants receive treatment for their colitis symptoms with one or more of several study drugs, which include mesalamine (5-ASA), corticosteroids, infliximab and 6-mercaptopurine, adalimumab and tacrolimus. The drugs are added to the treatment plan one at a time to find the combination that works best for the individual patient. Patients who respond to one or more of the medications may continue treatment with that same combination for up to 6 months.

Regular clinic visits are scheduled for blood tests, symptoms ratings questionnaires and periodic physical examinations and colonoscopies to measure the response to treatment and evaluate any side effects.

DETAILED DESCRIPTION:
The primary purpose of this study is to detect patterns of immune abnormalities in the colitis associated with Hermansky-Pudlak Syndrome (HPS). Additionally we aim to document the clinical response to and tolerance of conventional inflammatory bowel disease (IBD) therapy for HPS patients with active colitis associated with Hermansky-Pudlak Syndrome (HPS). HPS is a rare autosomal recessive disorder causing dysfunctional lysosome-related organelle formation and trafficking resulting in oculocutaneous albinism and a bleeding diathesis secondary to platelet dysfunction. Associated conditions include pulmonary fibrosis, IBD, and systemic ceroid deposition. The associated IBD has been reported to occur at a higher frequency in the HPS-1 and HPS-4 subtypes compared to the prevalence of IBD in non-HPS populations. HPS IBD has clinical features of both ulcerative colitis (UC) and Crohn's disease, but histologically resembles Crohn's disease in that granulomas are commonly seen in the mucosa of the intestine. The pathogenesis of HPS IBD is not fully understood and little data beyond descriptions of the clinical and histologic manifestations have been published. Furthermore reports on treatment of the colitis in HPS patients are largely anecdotal, and our own experience suggests that many patients may be under-treated.

HPS patients with active colitis will be enrolled into this prospective treatment study. Endpoints for the immunopathogenesis studies will include baseline measurements of and changes in immune cell populations, cytokine, and chemokine expression. In the blood and gut mucosa. Endpoints for the study of response to treatment will include changes in clinical, endoscopic, and histologic scores as well as the rate and severity of adverse events. Descriptive summary statistical analysis (n, mean, median, standard deviation, minimum and maximum range) and simple correlations of clinical response variables with immune parameters will be done.

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject is eligible for the study if all of the following criteria are met:

* Has given written informed consent prior to screening.
* Age 18 years old or greater.
* Has confirmed diagnosis of HPS prior to screening.
* Has confirmed diagnosis of IBD prior to screening.
* The presence of active disease as defined by a SCCAI score greater than or equal to 5.
* Negative results on stool examination for culture of enteric pathogens (Salmonella, Shigella, Yersinia, Campylobacter, Vibrio, E. coli O157/H7), Clostridium difficile toxin assay, enteric parasites and their ova (including Giardia and Cryptosporidia).
* If currently receiving medication for their IBD, patients may be on a stable regimen of one or a combination of the following drug doses and durations:

Corticosteroids (less than or equal to 25 milligrams Prednisone or Prednisone equivalent per day) - greater than or equal to 4 weeks.

5-ASA Sulfasalazine - greater than or equal to 4 weeks.

Azathioprine/6-MP/thioguanine with stable dose for eight weeks - greater than or equal to 12 weeks. (NOTE: Patients receiving azathioprine/6-MP/thioguanine must have been on a stable dose of this medication for greater than or equal to 8 weeks)

Probiotics (live bacterial dietary supplements) - greater than or equal to 4 weeks.

Prebiotics (dietary supplements to produce biologically active substances) - greater than or equal to 4 weeks.

Infliximab (5 to 10 mg/kg IV) - greater than 8 weeks or no response within 4 weeks of an induction dose of 3 infusions.

Adalimumab (40 to 80 mg subq) - greater than or equal to 4 weeks or no response within 2 weeks after induction dose of 2 injections.

EXCLUSION CRITERIA:

A subject is excluded from the study if any of the following criteria are met:

GENERAL CRITERIA:

* Has any clinically significant disease (e.g., renal, hepatic, neurological, cardiovascular, pulmonary, endocrinology, psychiatric, hematological, urologic, or other acute or chronic illness) that in the opinion of the investigator would make the subject an unsuitable candidate for this trial.
* Inability to meet any of the above inclusion criteria.
* Is a woman who has a positive serum pregnancy test or who is breast-feeding.
* Has any of the following clinical chemistry values:

  1. AST greater than 2.5 times the upper limit of normal (ULN).
  2. ALT greater than 2.5 times the ULN.
  3. Serum bilirubin greater than 1.5 times the ULN.
  4. Serum creatinine greater than 1.5 times the ULN.
  5. Alkaline phosphatase greater than 2.5 times the ULN.
* Has a hemoglobin level less than 8.0 g/dL or hematocrit less than 26 percent.
* Has a PT INR greater than 1.3 or a PTT greater than 3 seconds compared to control value.
* Has the following cell counts:

  1. Platelet count less than 80,000 or greater than 950,000.
  2. White blood cell count less than 1200.
  3. Neutrophil count less than 700.
* Has a current infection requiring intravenous antibiotics, a serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., pneumonia, septicemia).
* Has a history of cancer within the past 5 years, with the exception of excised basal cell carcinoma, squamous cell carcinoma of the skin, or cervical carcinoma in situ.
* Had a dependency for any illicit drug, chemical or alcohol within the past 5 years.
* Has a history of active tuberculosis (TB) (or a positive PPD skin test or chest x-ray with findings suggestive of old TB infection including calcified nodular lesions, apical fibrosis, or pleural scarring), acute or chronic hepatitis B, hepatitis C, human immunodeficiency virus (HIV).
* History of central nervous system demyelinating disease, or systemic lupus erythematosus.
* Unable to keep to the scheduled appointments and other test to watch for changes in symptoms and side effects of treatment.

GASTROINTESTINAL CRITERIA:

* History of colectomy, partial colectomy, current ostomy, pouchitis, or small bowel resection within the past 6 months, or short gut syndrome.
* Presence of current active bowel obstruction, intestinal perforation, known presence of high grade stricture, history of toxic megacolon, history of colonic epithelium high-grade dysplasia or a dysplasia-associated lesion or mass that does not resemble an adenoma (that is a mass lesion, stricture, or broad-based tumor with dysplasia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08-07; Primary Completion 2011-03-08 (Actual); Study Completion 2011-03-08 (Actual)

PRIMARY OUTCOMES:
To detect patterns of immune abnormalities in the colitis associated with Hermansky-Pudlak Syndrome (HPS). | 60 weeks

SECONDARY OUTCOMES:
Document the clinical response to and tolerance of conventional inflammatory bowel disease (IBD) therapy for HPS patients with active colitis associated with Hermansky-Pudlak Syndrome (HPS). | 60 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bergman R, Parkes M. Systematic review: the use of mesalazine in inflammatory bowel disease. Aliment Pharmacol Ther. 2006 Apr 1;23(7):841-55. doi: 10.1111/j.1365-2036.2006.02846.x. PMID 16573787
- [Background] Cappell MS. Gastrointestinal endoscopy in high-risk patients. Dig Dis. 1996 Jul-Aug;14(4):228-44. doi: 10.1159/000171555. PMID 8843979
- [Background] D'Haens G, Daperno M. Advances in biologic therapy for ulcerative colitis and Crohn's disease. Curr Gastroenterol Rep. 2006 Dec;8(6):506-12. doi: 10.1007/s11894-006-0041-5. PMID 17105690